CLINICAL TRIAL: NCT01248988
Title: Safety of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal-protein D-diphtheria Toxoid-tetanus Toxoid Conjugate (10PN-PD-DiT) Vaccine, Synflorix When Administered According to the Approved Prescribing Information in Korea
Brief Title: Post Marketing Surveillance of Synflorix Vaccine Safety Among Infants in Korea
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114469
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Safety; Synflorix; Pneumococcal diseases
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Synflorix Group: Infants and children who received at least one dose of Synflorix™ as a part of routine practice at a private clinic or hospital
  Interventions: Other: Synflorix™ Data collection

INTERVENTIONS:
Other: Synflorix™ Data collection — Safety monitoring: recording of adverse events during using diary cards and recording of serious adverse events using the latest version of Korea's Post-Marketing Surveillance Serious Adverse Event Reporting Form.

SUMMARY:
The purpose of this study is to collect safety information following routine vaccination with Synflorix™ among infants in Korea.

DETAILED DESCRIPTION:
Rationale for the protocol amendment: The therapeutic indication for Synflorix in Korea has been updated. The protocol is being amended to reflect this update.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representatives can and will comply with the requirements of the protocol.
* Korean male or female subjects whose age while receiving the first vaccination with Synflorix is 6 weeks - 5 years.
* Written, signed or thumb-printed informed consent obtained from the parent(s)/ Legally Acceptable Representative(s) of the child. Where parent(s)/Legally acceptable representatives are illiterate, the consent form will be countersigned by a witness.

Exclusion Criteria:

* At the time of Post Marketing Surveillance entry, the contraindications and precautions of use indicated in the local Prescribing Information should be checked and the infant must not be included in the Post Marketing Surveillance if there is any contraindication. Any changes in the locally approved Prescribing Information must be implemented immediately.
* Subjects who receive any investigational or non-registered pneumococcal vaccine 30 days prior to the study start will not be enrolled. Subjects who had previous administration of a pneumococcal vaccine other than Synforix will not be enrolled into the study.
* A male or female children >= 5 years of age at study entry.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children who receive at least one dose of Synflorix as a part of routine practice at a private clinic or hospital.
Sampling Method: Non-Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2010-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of unexpected adverse events | During the 30-day (Day 0 - Day 29) follow-up period after each vaccine dose.
Occurrence of expected adverse events | During the 30-day (Day 0 - Day 29) follow-up period after each vaccine dose.
Occurrence of serious adverse events | From the first dose in the study up to 30 days (Day 0 - Day 29) after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Suwon, Kyonggi-do, South Korea

REFERENCES:
- [Derived] Lee SM, Lee JH, Song ES, Kim SJ, Kim JH, Jakes RW, Devadiga R, Park MS. A 6-year safety surveillance of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in South Korea. Hum Vaccin Immunother. 2018;14(12):3019-3025. doi: 10.1080/21645515.2018.1502525. Epub 2018 Aug 29. PMID 30084702